CLINICAL TRIAL: NCT02805075
Title: Single Arm Dose-Escalation Trial of Fructo-Oligosaccharides in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Fructooligosaccharides in Treating Patients With Blood Cancer Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Rezvani, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BMT303; NCI-2016-00847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 37379 (Other: Stanford IRB); P30CA124435 (NIH)
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Recurrent Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fructooligosaccharide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (Fructooligosaccharide) (Experimental): Patients receive FOS PO BID for 21 days starting at 7 days before allogeneic hematopoietic stem cell transplant in the absence of disease progression or unexpected toxicity.
  Interventions: Other: Fructooligosaccharide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Fructooligosaccharide — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies the side effects and best dose of fructooligosaccharides in treating patients with blood cancer who are undergoing donor stem cell transplant. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Nutritional supplements such as fructooligosaccharides may reduce the incidence of graft-versus-host disease in patients with blood cancer undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a dose escalation trial to determine the tolerability of the fructo-oligosaccharides prebiotic in allogeneic hematopoeitic stem cell transplant (HSCT) patients.

OUTLINE: This is a dose escalation study.

Patients receive fructooligosaccharides (FOS) orally (PO) twice daily (BID) for 21 days starting at 7 days before allogeneic hematopoietic stem cell transplant in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study will have a hematologic malignancy (any stage or grade) for which they are undergoing preparation for allogeneic HSCT; participants in the study will be restricted to those undergoing HSCT under reduced-intensity protocols 9924 and 9907
* No limitations exist for type or amount of prior therapy
* No restrictions or requirements will be placed on race
* No restrictions will be made based on life expectancy
* Patients will not be evaluated based on Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status (KPS)
* No restrictions will be made based on organ or marrow function
* Patients will be included only if they have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a history of gastric bypass surgery or inflammatory bowel disease
* Patients with a history of or current bowel obstruction
* Patients actively enrolled on any other GVHD prevention trial
* Patients with known fructose intolerance
* Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient or raise concern that the patient would not comply with protocol procedures
* Subjects may co-enroll on other investigational studies except for investigational studies whose primary aim is the prevention of GVHD
* No additional restrictions exist regarding co-morbid disease or incurrent illness
* Patients will be excluded from the trial if they have had a history of allergies or intolerance to fructooligosaccharides or the components of FOS including fructose and glucose
* No exclusion is necessary based on the use of other concomitant medications; specifically there is no prohibition of concomitant antibiotic, antiviral or antifungal therapy; subjects may co-enroll on other investigational studies except for investigational studies whose primary aim is the prevention of GVHD
* Pregnant or nursing patients will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the ability to take 70% of all doses over 21 days | At day 21
  Will employ the Bayesian optimal interval design.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rezvani, Principal Investigator — Stanford University; Tessa Andermann, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States